## ID: 170577

## Management of Severe Acute Malnutrition in SCD, in Northern Nigeria

NCT03634488

Protocol Version: 06/01/2022

## Statistical Analysis

Data was collected and managed with Research Electronic Data Capture (REDCap) hosted at Vanderbilt University Medical Center. We summarized continuous variables as means and standard deviations (sd) or as medians and interquartile ranges (IQR) for variables not normally distributed. Categorical variables and prevalence were reported as numbers and percentages. For comparisons between groups, a chi-square test or Fisher's exact test was used for percentages, a t-test for means, and a Mann-Whitney U test for medians.

We used two regression models to study characteristics associated with weight gain for all participants with SCD. Per protocol, we used a logistic regression model to study whether participants achieved a BMI z-score of at least -3.0 and whether they achieved at least a 15% weight gain. Finally, due to the evidence that weight-for-age z-score is associated with mortality in children with SCA in the same age range living in northern Nigeria, we utilized the same covariates for the logistic mode for a linear regression model to study the change in weight-forage z-score from baseline.

1. Klein LJ, Abdullahi SU, Gambo S, et al. Underweight children older than 5 years with sickle cell anemia are at risk for early mortality in a low-resource setting. *Blood Adv.* 2023;7(11):2339-2346.